CLINICAL TRIAL: NCT00993499
Title: A Phase Ib Open Label Clinical Trial of Continuous Once Daily Oral Treatment Using BIBW 2992 Plus Sirolimus in Patients With Non-small Cell Lung Cancer Harbouring an EGFR Mutation and/or Disease Progression Following Prior Erlotinib or Gefitinib
Brief Title: Trial of Continuous Once Daily Oral Treatment Using BIBW 2992 (Afatinib) Plus Sirolimus (Rapamune®) in Patients With Non-small Cell Lung Cancer Harbouring an EGFR Mutation and/or Disease Progression Following Prior Erlotinib or Gefitinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.70; 2009-010432-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Sirolimus

ARMS (1):
- BIBW 2992 + Sirolimus (Experimental): Dose escalation of the combination BIBW 2992 plus Sirolimus.
  Interventions: Drug: BIBW 2992; Drug: Sirolimus (rapamycin)

INTERVENTIONS:
Drug: BIBW 2992 — Dose escalation (19-40 patients): low or high dose oral + 12 addit. pat. at MTD, until progression or undue AEs
Drug: Sirolimus (rapamycin) — Dose escalation (19-40 patients): several dose levels + 12 addit. pat. at MTD until progression or undue AEs.

SUMMARY:
The primary objective of this trial is to identify the Maximum Tolerated Dose of BIBW 2992 therapy when given continuously in combination with Sirolimus.

The MTD will be based on the Dose Limiting Toxicity information collected during the first two cycles.

Overall safety, pharmacokinetics and anti-tumour efficacy will be evaluated as secondary objectives.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically or cytologically confirmed diagnosis of Stage IIIB or Stage IV NSCLC
2. Patients who have failed conventional treatment (at least 1 prior treatment line), or for whom no therapy of proven efficacy exists
3. Patients whose tumors:

   * are EGFR mutation-positive or
   * are EGFR mutation-negative or unknown provided they had disease progression after achieving either response or stable disease for at least 6 months from a previous treatment with erlotinib (Tarceva®) or gefitinib (Iressa®)
4. Patients aged 18 years or older
5. Life expectancy of at least three (3) months
6. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score 0-2
7. Written informed consent that is consistent with ICH-GCP guidelines

Exclusion criteria:

1. Prior major surgery, chemotherapy or radiation therapy within 4 weeks before start of therapy.
2. Prior treatment with an mTOR inhibitor within the past 4 weeks before start of therapy or concomitantly with this study
3. Use of erlotinib (Tarceva®) or gefitinib (Iressa®) within 14 days of run-in treatment with Sirolimus
4. Active CNS metastases (defined as stable for <4 weeks and/or symptomatic and/or requiring treatment with anticonvulsants or steroids)
5. Severe alteration in serum fasting cholesterol (equal or more than 350 mg/dL) or triglycerides (equal or more than 400 mg/dL). Patients may be allowed to enrol on the trial after initiation of lipid lowering agents.
6. Requirement for treatment with any of the prohibited concomitant medications:

   * Concomitant CYP3A4 inhibitors within the past 7 days before start of therapy or concomitantly with this study.
   * Concomitant CYP3A4 inducers within the past 14 days before start of therapy or concomitantly with this study.
7. Any contraindications for therapy with Sirolimus.
8. Known hypersensitivity to BIBW 2992, Sirolimus or other rapamycin analogues (everolimus, temsirolimus, deforolimus, etc.) or the excipients of any of the trial drugs.
9. Use of any investigational drug within 4 weeks before start of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (8):
- Spain (8):
  - 1200.70.34001 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 1200.70.34008 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.70.34009 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.70.34006 Boehringer Ingelheim Investigational Site, Girona
  - 1200.70.34007 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1200.70.34005 Boehringer Ingelheim Investigational Site, Majadahonda (Madrid)
  - 1200.70.34004 Boehringer Ingelheim Investigational Site, Valencia
  - 1200.70.34002 Boehringer Ingelheim Investigational Site, Zaragoza

REFERENCES:
- [Derived] Moran T, Palmero R, Provencio M, Insa A, Majem M, Reguart N, Bosch-Barrera J, Isla D, Costa EC, Lee C, Puig M, Kraemer S, Schnell D, Rosell R. A phase Ib trial of continuous once-daily oral afatinib plus sirolimus in patients with epidermal growth factor receptor mutation-positive non-small cell lung cancer and/or disease progression following prior erlotinib or gefitinib. Lung Cancer. 2017 Jun;108:154-160. doi: 10.1016/j.lungcan.2017.03.009. Epub 2017 Mar 22. PMID 28625629

RESULTS

PARTICIPANT FLOW:
Groups:
- Afa30+Sir01: Patients received Sirolimus (Sir) 1mg tablet orally for 8 days, followed by oral administration of Afatinib (Afa) 30mg tablet once daily plus Sir 1mg tablet once daily.
- Afa30+Sir03: Patients received Sirolimus (Sir) 1mg tablet orally for 8 days, followed by oral administration of Afatinib (Afa) 30mg tablet once daily plus Sir 3mg tablet once daily.
- Afa30+Sir05: Patients received Sirolimus (Sir) 1mg tablet orally for 8 days, followed by oral administration of Afatinib (Afa) 30mg tablet once daily plus Sir 5mg tablet once daily.
- Afa30+Sir10: Patients received Sirolimus (Sir) 1mg tablet orally for 8 days, followed by oral administration of Afatinib (Afa) 30mg tablet once daily plus Sir 10mg tablet once daily.
- Afa40+Sir01: Patients received Sirolimus (Sir) 1mg tablet orally for 8 days, followed by oral administration of Afatinib (Afa) 40mg tablet once daily plus Sir 1mg tablet once daily.
- Afa40+Sir05: Patients received Sirolimus (Sir) 1mg tablet orally for 8 days, followed by oral administration of Afatinib (Afa) 40mg tablet once daily plus Sir 5mg tablet once daily.
Period: Run-in Period (8 Days)
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Started | 13 | 12 | 10 | 3 | 3 | 3
Completed | 12 | 9 | 9 | 3 | 3 | 3
Not Completed | 1 | 3 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Inclusion/exclusion criteria not met | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 1 | 0 | 0 | 0
Period: Discontinued Before Starting Course 3
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Started | 12 | 9 | 9 | 3 | 3 | 3
Completed | 8 | 5 | 6 | 2 | 3 | 3
Not Completed | 4 | 4 | 3 | 1 | 0 | 0
Not completed — Progressive Disease | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Dose Limiting Toxicity (DLT) | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Non compliance with the protocol | 0 | 0 | 2 | 0 | 0 | 0
Period: Discontinued After Starting Course 3
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Started | 12 | 9 | 9 | 3 | 3 | 3
Completed | 4 | 4 | 3 | 1 | 0 | 0
Not Completed | 8 | 5 | 6 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 6 | 4 | 3 | 1 | 3 | 3
Not completed — DLT | 1 | 0 | 2 | 1 | 0 | 0
Not completed — Other adverse event | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who recieved at least one dose of the trial drug during the first and second treatment counrses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05 | Total
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (13.6) | 56.5 (12.5) | 65.1 (9.6) | 50.8 (7.5) | 53.4 (12.4) | 56.5 (17.2) | 58.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 4 | 1 | 2 | 2 | 24
  Male | 3 | 3 | 5 | 2 | 1 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Dose Limiting Toxicities (DLT)
Description: Number of participants with of dose limiting toxicities (DLT)
Time Frame: 2 first cycles, 56 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Participants | 3 | 2 | 4 | 3 | 2 | 3

2. Secondary Outcome: Best Overall Response
Description: Best overall response (unconfirmed) according to RECIST v1.1
Time Frame: From first trial medication intake in the first treatment course until last trial medication intake plus 28 days, up to 367 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Percentage of participants
  Complete Response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Partial Response | 8.3 | 0.0 | 22.2 | 0.0 | 0.0 | 66.7
  Stable Disease | 50.0 | 44.4 | 44.4 | 33.3 | 66.7 | 33.3
  Progressive Disease | 33.3 | 22.2 | 11.1 | 33.3 | 33.3 | 0.0
  Not evaluable | 8.3 | 0.0 | 11.1 | 33.3 | 0.0 | 0.0
  Missing (baseline data only) | 0.0 | 33.3 | 11.1 | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Objective Response
Description: Rate of (unconfirmed) objective response, defined as complete response (CR) or partial response (PR) according to RECIST v1.1
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Percentage of participants | 8.3 | 0.0 | 22.2 | 0.0 | 0.0 | 66.7

4. Secondary Outcome: Rate of Disease Control
Description: Rate of (unconfirmed) disease control defined as CR, PR, or stable disease (SD), according to RECIST v1.1
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Percentage of participants | 58.3 | 44.4 | 66.7 | 33.3 | 66.7 | 100.0

5. Secondary Outcome: Exploratory Examination of EGFR Mutations (Exons 19, 20 and 21 and Others) in Serum/Plasma DNA and Tumour DNA.
Description: Exploratory examination of Epidermal growth factor (receptor)(EGFR) mutations (Exons 19, 20 and 21 and others) in serum/plasma DNA and tumour DNA.
  This endpoint was not analysed in the study report as the available data was too limited.
Time Frame: Multiple time points during the trial
Population: Treated set. This endpoint was not analysed in the study report as the available data was too limited.
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Measured Plasma Concentration of Afatinib at Steady State (Cmax,ss)
Description: Maximum measured plasma concentration of Afatinib at steady state (Cmax,ss)
Time Frame: 24 hours (h), 311h 55minutes (min), 312h, 313h, 314h, 315h, 316h, 317h, 318h, 320h and 336h after first administration of afatinib
Population: Pharmacokinetic (PK) set which included all patients in the treated set who had taken at least 1 dose of study medication and for whom at least 1 valid blood or plasma concentration was available. No patients in the Afa40+Sir05 group had analyzable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 7 | 6 | 3 | 2 | 2 | 0
ng/mL | 41.4 (17.6) | 47.1 (63.8) | 98.1 (33.9) | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. |

7. Secondary Outcome: AUC of Afatinib at Steady State Over the Dosing Interval τ (AUCτ,ss)
Description: Area under the curve (AUC) of Afatinib at steady state over the dosing interval τ (AUCτ,ss) for afatinib.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 6 | 4 | 3 | 2 | 1 | 0
ng*h/mL | 603 (37.3) | 536 (40.1) | 1560 (49.6) | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | 1760 (NA) — Not calculable as only one patient with data. |

8. Secondary Outcome: Maximum Measured Plasma Concentration of Sirolimus at Steady State (Cmax,ss)
Description: Maximum measured plasma concentration of sirolimus at steady state (Cmax,ss)
Time Frame: 24 hours (h) 5 minutes (min), 24h, 23h, 22h, 20h, 18h, 16h, 5min before first afatinib administration and 144h, 311h 55min, 312h, 313h, 314h, 315h, 316h, 317h, 318h, 320h, 336h, 480h after first administration of afatinib
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 8 | 5 | 7 | 2 | 2 | 3
ng/mL
  Sirolimus alone (N=8, 5, 7, 1, 2, 3) | 7.96 (40.7) | 13.8 (24.1) | 32.5 (43.8) | 30.2 (NA) — Not calculable as only one patient with data. | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | 28.5 (21.9)
  Sirolimus with Afatinib (N=6, 3, 2, 2, 1, 0) | 5.81 (64.6) | 15.3 (1.31) | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | 8.53 (NA) — Not calculable as only one patient with data. | NA (NA) — No patients with analyzable data

9. Secondary Outcome: AUC of Sirolimus at Steady State Over the Dosing Interval τ (AUCτ,ss)
Description: Area under the curve (AUC) of sirolimus at steady state over the dosing interval τ (AUCτ,ss) for afatinib.
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 6 | 4 | 7 | 2 | 2 | 2
ng*h/mL
  Sirolimus alone (N=6, 4, 7, 1, 2, 2) | 91.5 (28.1) | 193 (35.4) | 502 (51.7) | 497 (NA) — Not calculable as only one patient with data. | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained.
  Sirolimus with Afatinib (N=4, 3, 2, 2, 1, 0) | 106 (57.9) | 207 (24.4) | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | NA (NA) — Not calculated as only 2 patients had data therefore a reliable estimate cannot be obtained. | 141 (NA) — Not calculable as only one patient with data. | NA (NA) — No patients with analyzable data

10. Secondary Outcome: Occurrence of Adverse Events According to CTCAE, Version 3.0
Description: Percentage of participants with adverse events according to highest Common Terminology Criteria for Adverse Events (CTCAE) grade, version 3.0
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Percentage of participants
  Grade 1 | 0.0 | 22.2 | 11.1 | 0.0 | 0.0 | 0.0
  Grade 2 | 33.3 | 0.0 | 22.2 | 0.0 | 0.0 | 0.0
  Grade 3 | 58.3 | 55.6 | 66.7 | 100.0 | 66.7 | 100.0
  Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0
  Grade 5 | 8.3 | 22.2 | 0.0 | 0.0 | 0.0 | 0.0

11. Secondary Outcome: Percentage of Patients With Drug-related AEs
Description: Percentage of patients with drug-related adverse events (AEs).
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

12. Secondary Outcome: Frequency of Patients With Possible Clinically-significant Abnormalities in Liver Enzymes or Total Bilirubin
Description: Evaluation of laboratory parameters included assessment of the frequency of patients with ALT and AST elevations concurrent with elevated bilirubin and indicative of Hy's law cases.
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Number analyzed (Participants) | 12 | 9 | 9 | 3 | 3 | 3
Percentage of participants
  High AST (Aspartate aminotransferase) | 16.7 | 11.1 | 11.1 | 0.0 | 33.3 | 0.0
  High ALT (Alanine aminotransferase) | 16.7 | 11.1 | 22.2 | 0.0 | 0.0 | 0.0
  High alkaline phosphatase | 9.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  High total bilirubin | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first trial medication intake in the first treatment course until last trial medication intake plus 28 days, up to 367 days
Arm/Group | Afa30+Sir01 | Afa30+Sir03 | Afa30+Sir05 | Afa30+Sir10 | Afa40+Sir01 | Afa40+Sir05
Serious Adverse Events (participants affected / at risk) | 4/12 | 6/9 | 7/9 | 2/3 | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 12/12 | 9/9 | 8/9 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afa30+Sir01 (N=12) | Afa30+Sir03 (N=9) | Afa30+Sir05 (N=9) | Afa30+Sir10 (N=3) | Afa40+Sir01 (N=3) | Afa40+Sir05 (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 3 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afa30+Sir01 (N=12) | Afa30+Sir03 (N=9) | Afa30+Sir05 (N=9) | Afa30+Sir10 (N=3) | Afa40+Sir01 (N=3) | Afa40+Sir05 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Trichomegaly (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 7 | 7 | 3 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 5 | 1 | 2 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1 | 2
Tooth discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4 | 1 | 1 | 0
Asthenia (General disorders) | 7 | 3 | 4 | 2 | 2 | 2
Chest pain (General disorders) | 2 | 0 | 1 | 0 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 5 | 6 | 4 | 3 | 1 | 2
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 2 | 1 | 1 | 2
Xerosis (General disorders) | 3 | 0 | 2 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 2 | 1 | 2 | 0 | 1 | 1
Periumbilical abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1 | 0 | 3 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 4 | 3 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Alexia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 5 | 4 | 2 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.